CLINICAL TRIAL: NCT05620979
Title: Evaluating the Role of Financial Navigation in Alleviating Financial Distress Among Young Adult Survivors of Blood Cancer
Brief Title: Financial Navigation Study Among Young Adult Blood Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts Medical Center (Other)
Collaborators: The Leukemia and Lymphoma Society (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY00001828
Record Dates: First submitted 2022-10-31; First posted 2022-11-17 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Survivorship; Cancer; Financial Stress
MeSH Terms: conditions — Neoplasms; Financial Stress

STUDY DESIGN:
Intervention Model Description: This is a multi-site, three-arm, financial navigation intervention
Masking Description: no blinding
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Active Navigation (Active Comparator): Active navigation with the study-based financial navigator scheduling four check-in meetings throughout the study with the participant. All participants will complete an assessment at baseline, 3 months and 6 months and be invited to participate in an optional interview after the 6-month assessment.
  Interventions: Behavioral: Providing financial navigation via active navigation, ad hoc navigation or no study-based navigation.
- Ad Hoc Navigation (Active Comparator): Ad hoc navigation in which participant is provided study-based financial navigator to contact as needed. All participants will complete an assessment at baseline, 3 months and 6 months and be invited to participate in an optional interview after the 6-month assessment.
  Interventions: Behavioral: Providing financial navigation via active navigation, ad hoc navigation or no study-based navigation.
- No study-based Navigation (Active Comparator): No access to a study-based financial navigator, but access to a national hotline through the Leukemia & Lymphoma Society. All participants will complete an assessment at baseline, 3 months and 6 months and be invited to participate in an optional interview after the 6-month assessment.
  Interventions: Behavioral: Providing financial navigation via active navigation, ad hoc navigation or no study-based navigation.

INTERVENTIONS:
Behavioral: Providing financial navigation via active navigation, ad hoc navigation or no study-based navigation. — Providing financial navigation to blood cancer survivors.

SUMMARY:
Young adult cancer survivors (18-39y) are at increased risk of financial distress. This study seeks to better understand the financial challenges experienced by these individuals via quantitative serial assessments, study-based financial navigator encounters and an end of study qualitative interview.

DETAILED DESCRIPTION:
This fully remote, multi-site study will evaluate the role of financial navigators in relieving financial distress in young adults (18-39y) who have completed treatment for blood cancer at least three years ago. Serial Assessments at study entry, 3-months, and 6-months measure financial distress measured using the study's primary outcome measure the Personal Financial Wellness Scale™ (PFW) (see below), hypothesized effect modifiers (emotional distress, self-efficacy, cognitive functioning), as well as care seeking, household finances and insurance characteristics. Randomization will occur following completion of baseline measures (see below for description of study arms). In addition to a formal evaluation of the intervention at 3- and 6-months, an optional interview will occur following the 6-month assessment/navigation intervention period to gain further insight from participants about the acceptability of the intervention. For ethical considerations related to the topic of study, all participants will be provided with the Leukemia & Lymphoma Society's information specialist hotline.

ELIGIBILITY:
Inclusion Criteria:

1. Previous diagnosis and treatment of blood cancer (leukemia, lymphoma, myeloma, myelodysplastic syndrome, or myeloproliferative neoplasm)
2. Current age between 18-39 years old
3. Blood cancer diagnosis during childhood (0-17 years of age) or young adulthood (18-36 years of age)
4. At least three years post blood cancer diagnosis
5. Off treatment for blood cancer or on a long-term regimen with an oral anti-cancer medication with stable disease
6. Off treatment for a second cancer (non-blood cancer) or on a stable long-term regimen, such as hormone therapy or hormone replacement therapy
7. Primary residence in United States
8. Able to understand and read the English language

Exclusion Criteria:

* On parent or guardian's insurance

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 130 (Actual)
Dates: Start 2022-02-14 (Actual); Primary Completion 2023-11-06 (Actual); Study Completion 2023-11-23 (Actual)

PRIMARY OUTCOMES:
Personal Financial Wellness Scale (PFW) | 6 months
  To evaluate the change in financial distress associated with randomization group assignment from baseline to 6-month follow up as measured by the 8-item Personal Financial Wellness Scale (PFW). The PFW scores range from 1-10 where lower scores indicate greater financial distress.

SECONDARY OUTCOMES:
Health-Related Quality of Life (HrQoL) Measures | 6 months
  As part of Aim 1, we will explore whether changes in financial distress (baseline to 6-months) are moderated by emotional distress, self-efficacy, and cognitive functioning, as measured by Patient-Reported Measurement Information System (PROMIS) 4-item short forms for emotions distress (depression and anxiety) and self-efficacy, as well as the 4-item cognitive functioning scale from the Quality of Life in Neurological Disorders (Neuro-Qol) battery. For each of these short forms, high scores connote better functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Susan K Parsons, MD, MRP, Principal Investigator — Tufts Medical Center
Locations (5):
- United States (5):
  - Children's Hospital Los Angeles, Los Angeles, California
  - University of Southern California (USC Norris Comprehensive Cancer Center & LA County Hospital), Los Angeles, California
  - Tufts Medical Center, Boston, Massachusetts
  - Bon Secours Mercy Health System, Greenville, South Carolina
  - MD Anderson, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ohlsen TJD, Murphy-Banks R, Beauchemin MP, Rodday AM, Freyer DR, Miller KA, Fleisher E, Xiang Q, Linendoll N, Chan RY, Crosswell HE, Roth ME, Parsons SK. Cancer-Related Impacts on Employment and Strategies for Support Among Long-Term Young Adult Survivors of Hematologic Malignancies. JCO Oncol Pract. 2025 Dec 12:OP2500558. doi: 10.1200/OP-25-00558. Online ahead of print. PMID 41385752
- [Derived] Beauchemin MP, Murphy-Banks R, Rodday AM, Freyer DR, Miller KA, Fleisher E, Ohlsen TJD, Linendoll N, Chan RY, Crosswell HE, Roth ME, Parsons SK. Factors influencing engagement in survivorship care among young adult survivors of hematologic malignancies: a mixed methods report. Support Care Cancer. 2025 Jun 25;33(7):628. doi: 10.1007/s00520-025-09686-1. PMID 40562962
- [Derived] Zheng DJ, Murphy-Banks R, Rodday AM, Xiang Q, Linendoll N, Beauchemin M, Ohlsen TJD, Fleisher E, Miller KA, Freyer DR, Crosswell HE, Chan RY, Roth ME, Parsons SK. "Nothing Is as Great a Learning Experience as Getting a $15,000 Bill": A Mixed-Methods Study of Young Adult Cancer Survivors' Experience With Insurance Coverage. JCO Oncol Pract. 2025 Jun 16:OP2401075. doi: 10.1200/OP-24-01075. Online ahead of print. PMID 40523211
- [Derived] Parsons SK, Murphy-Banks R, Rodday AM, Roth ME, Miller K, Linendoll N, Chan R, Crosswell HE, Xiang Q, Freyer DR. Financial distress and medical financial hardship among young adult survivors of blood cancer. JNCI Cancer Spectr. 2024 Sep 2;8(5):pkae071. doi: 10.1093/jncics/pkae071. PMID 39153000